## A novel estimation of energy balance through the calibration of consumer devices in free-living, US adults and children

Statistical Analysis Plan

1/9/2018

## Statistical Analyses

Statistical significance for comparison between the different data collection methodologies will be tested using analysis of variance (ANOVA) for continuous variables and chi-square tests for categorical variables. Statistical significance will be set at P<.05 (two-sided) for all analyses.